CLINICAL TRIAL: NCT01988805
Title: Immunological Characterization of Blood and Inflammasome Gene Segment Polymorphism Analysis of Normal Healthy Individuals
Brief Title: Gene Polymorphism Study of Normal Individual Inflammasome Genes
Status: Withdrawn | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Mark D. Wewers, MD, Associate Director, Pulmonary Research, Ohio State University
Other Study IDs: 2012H0346
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Individuals
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Blood Draw: Normal healthy individuals will be consented and their blood drawn at the time of their visit.
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw

SUMMARY:
This study is intended to collect blood from healthy individuals to investigate whether variations in immune-related (inflammasome) genes affect how the immune cells found in the blood can help fight infections and prevent diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy with no chronic or acute illnesses, or taking medication which in the opinion of the PI would impact the analyses being conducted.
2. At least 18 years or older.
3. Are capable of reading, understanding and providing written informed consent.

Exclusion Criteria:

1. Non-English speaking.
2. Individuals under 18 years old.
3. Woman who believe they are or may be pregnant. (Based on self reporting. Pregnancy testing will not be conducted for the purposes of this study)
4. Individuals experiencing acute or chronic illnesses which in the opinion of the PI would impact the analyses being conducted.
5. Currently taking prescription or over the counter medication which in the opinion of the PI would impact the analyses being conducted.
6. Individual has donated blood more than twice in the last week or the amount to be drawn will exceed the maximum allowance in the last 8 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
analyze their ability to respond to exogenous challenges by changing the production of proteins, the expression of genes and their ability to migrate and ingest materials | one visit
  Our intent is to collect these cells, divide them into subtypes such as monocytes, lymphocytes and neutrophils and then to analyze their ability to respond to exogenous challenges by changing the production of proteins, the expression of genes and their ability to migrate and ingest materials. We additionally will be interested in examining the cell components that may be released from these cells during various in vitro challenges.

CONTACTS AND LOCATIONS:
Locations (1):
- Davis Heart & Lung Research Institute, Columbus, Ohio, United States